CLINICAL TRIAL: NCT02581189
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Canada (AMBER)
Brief Title: Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C in Canada
Acronym: AMBER
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Collaborators: IST GmbH, Germany (Industry); Cato Research (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-651
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Effectiveness; Influence of adherence; Patient reported outcomes; Ombitasvir/paritaprevir/ritonavir ± dasabuvir; Chronic Hepatitis C genotype 1; Chronic Hepatitis C genotype 4
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — ombitasvir; paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with HCV genotype 1 or 4: Ombitasvir/paritaprevir/ritonavir (two 12.5 mg/75 mg/50 mg co-formulated tablets once daily); ± dasabuvir (tablet; 250 mg twice daily); ± weight-based ribavirin (tablet; 1000 or 1200 mg divided twice a day) up to 24 weeks
  Interventions: Drug: Ombitasvir/paritaprevir/ritonavir; Drug: Dasabuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Ombitasvir/paritaprevir/ritonavir — Co-formulated tablet
  Other Names: Ombitasvir also known as ABT-267; Paritaprevir also known as ABT-450
Drug: Dasabuvir — Tablet
  Other Names: ABT-333
Drug: Ribavirin — Tablet

SUMMARY:
The interferon-free combination regimen of ombitasvir/paritaprevir/ritonavir/ with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) for the treatment of chronic hepatitis C (CHC) has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well-controlled conditions. This observational study was the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in Canada in a clinical practice patient population.

DETAILED DESCRIPTION:
This was a prospective, multi-center observational study in participants receiving the interferon-free ABBVIE REGIMEN ± RBV in Canada. The prescription of a treatment regimen was at the discretion of the physician in accordance with local clinical practice and label, was made independently from this observational study and preceded the decision to offer the participant the opportunity to participate in this study. Adults chronically infected with HCV, receiving the interferon-free ABBVIE REGIMEN, were offered the opportunity to participate in this study during a routine clinical visit at the participating sites. Follow-up visits, treatment, procedures, and diagnostic methods followed physicians' routine clinical practice. Data were collected at the following time windows: baseline, early on-treatment visit, mid-treatment visit (for participants with a treatment duration of 24 weeks), end of treatment (EoT), early post-treatment and 12 and 24 weeks after the end of treatment (representing sustained virologic response 12 weeks after the end of treatment [SVR12] and sustained virologic response 24 weeks after the end of treatment [SVR24]).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced adult male or female participants with confirmed chronic hepatitis C (CHC), genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± ribavirin (RBV) according to standard of care and in line with the current local label
* If RBV was co-administered with the ABBVIE REGIMEN, it had to be prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)
* Participants had to voluntarily sign and date an informed consent form prior to inclusion into the study
* Participants must not have participated or intended to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic hepatitis C virus infection, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± ribavirin.
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Safety population: all enrolled participants receiving at least 1 dose of the ABBVIE REGIMEN.The prescribed ABBVIE REGIMEN needed to be known. 565 participants enrolled; treatment not started in 28 participants; 3 withdrew consent and no start of treatment was recorded; Two of the 3 deaths noted below occurred during the SAE collection period.
Period: Overall Study
Arm/Group | Participants With HCV Genotype 1 or 4
Started | 534
Completed | 481
Not Completed | 53
Not completed — Failure to return | 36
Not completed — Withdrew consent | 5
Not completed — Death | 3
Not completed — Insufficient virological response | 2
Not completed — Other, not specified | 7

BASELINE CHARACTERISTICS:
Population: Safety population: all enrolled participants who received at least one dose of the ABBVIE REGIMEN. The prescribed ABBVIE REGIMEN needed to be known.
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 534
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179
  Male | 355
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 426
  More than one race | 0
  Unknown or Not Reported | 35
Hepatitis C genotype [Count of Participants; unit: Participants]
  Genotype 1a | 286
  Genotype 1b | 221
  Genotype 4 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than 50 IU/mL 12 weeks after the last actual dose of study drug. The core population (CP) consisted of participants who met all inclusion criteria and were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype). The core population with sufficient follow-up data 12 weeks after the last actual dose of study drug (CPSFU12) was defined as all CP participants who fulfilled one of the following criteria:
  * evaluable HCV RNA data ≥70 days after the last actual dose of the ABBVIE REGIMEN
  * an HCV RNA value ≥50 IU/mL at the last measurement post-baseline
  * HCV RNA <50 IU/mL at the last measurement post-baseline, but no HCV RNA measurement ≥70 days after the last actual dose of the ABBVIE REGIMEN due to reasons related to safety (e.g. dropped out due to AE) or virologic failure
Time Frame: 12 weeks after the last actual dose of study drug
Population: Core population (CP) and core population with sufficient follow-up data 12 weeks after the last actual dose of study drug (CPSFU12) are defined in the outcome measure description
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants
  Core population (CP) | 86.6 [83.5 to 89.3]
  CPSFU12: number analyzed (Participants) | 489
  CPSFU12 | 94.1 [91.6 to 95.8]

2. Secondary Outcome: Percentage of Participants With Virologic Response at End of Treatment (EoT)
Description: Virologic response was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than 50 IU/mL at the end of treatment.
Time Frame: Up to 24 weeks
Population: Core population: Participants meeting all inclusion criteria and who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 93.8 [91.4 to 95.5]

3. Secondary Outcome: Percentage of Participants With Relapse
Description: Relapse was defined as hepatitis C virus ribonucleic acid (HCV RNA) level less than 50 IU/mL at the end of treatment followed by HCV RNA level greater than or equal to 50 IU/mL.
Time Frame: Up to 48 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 2.6 [1.5 to 4.5]

4. Secondary Outcome: Percentage of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as at least 1 documented hepatitis C virus ribonucleic acid (HCV RNA) level less than 50 IU/mL followed by HCV RNA level greater than or equal to 50 IU/mL during treatment.
Time Frame: Up to 24 weeks
Population: Core population (those meeting inclusion criteria and treated according to the standard of care and w/in local label guidelines for specific disease characteristics [cirrhotic status, genotype]) who had at least 1 undetectable or unquantifiable, on-treatment HCV RNA measurement and at least 1 on-treatment or end of treatment measurement thereafter
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 0.9 [0.3 to 3.4]

5. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as breakthrough (at least 1 documented hepatitis C virus ribonucleic acid (HCV RNA) less than 50 IU/mL followed by HCV RNA greater than or equal to 50 IU/mL during treatment) or failure to suppress (each measured on-treatment HCV RNA value greater than or equal to 50 IU/mL).
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 1.3

6. Secondary Outcome: Percentage of Participants Meeting Relapse Criteria
Description: Relapse was defined as hepatitis C virus ribonucleic acid (HCV RNA) less than 50 IU/mL at end of treatment or at the last on-treatment HCV RNA measurement followed by HCV RNA greater than or equal to 50 IU/mL post-treatment.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 2.1

7. Secondary Outcome: Percentage of Participants Meeting Premature Study Drug Discontinuation Criteria
Description: Premature study drug discontinuation was defined as participants who prematurely discontinued study drug with no on-treatment virologic failure.
Time Frame: 12 weeks after the last actual dose of study drug
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 2.1

8. Secondary Outcome: Percentage of Participants With Missing Sustained Virologic Response 12 Weeks Post-Treatment (SVR12) Data and/or Nonresponders Who Did Not Meet Specific SVR12 Nonresponder Criteria
Description: The number of participants with missing SVR12 data or SVR12 nonresponder participants who did not meet criteria for on-treatment virologic failure, relapse, premature treatment discontinuation, and who did not have an Insufficient virological response reported was documented.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Participants meeting all inclusion criteria and who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype)
Measure: Number; unit: percentage of participants
Arm/Group | Participants With HCV Genotype 1 or 4
Number analyzed (Participants) | 531
percentage of participants | 6.6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.Two of the 3 deaths noted below occurred during the SAE collection period.
Groups:
- Ombitasvir/Paritaprevir/Ritonavir: Ombitasvir/paritaprevir/ritonavir (two 12.5 mg/75 mg/50 mg co-formulated tablets once daily) up to 24 weeks
- Ombitasvir/Paritaprevir/Ritonavir + Ribavirin: Ombitasvir/paritaprevir/ritonavir (two 12.5 mg/75 mg/50 mg co-formulated tablets once daily) + weight-based ribavirin (tablet; 1000 or 1200 mg divided twice a day) up to 24 weeks
- Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir: Ombitasvir/paritaprevir/ritonavir (two 12.5 mg/75 mg/50 mg co-formulated tablets once daily) + dasabuvir (tablet; 250 mg twice daily) up to 24 weeks
- Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + Ribavirin: Ombitasvir/paritaprevir/ritonavir (two 12.5 mg/75 mg/50 mg co-formulated tablets once daily) + dasabuvir (tablet; 250 mg twice daily); + weight-based ribavirin (tablet; 1000 or 1200 mg divided twice a day) up to 24 weeks
Arm/Group | Ombitasvir/Paritaprevir/Ritonavir | Ombitasvir/Paritaprevir/Ritonavir + Ribavirin | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + Ribavirin
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/26 | 2/210 | 1/297
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/26 | 9/210 | 15/297
Other Adverse Events (participants affected / at risk) | 0/1 | 10/26 | 31/210 | 102/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir (N=1) | Ombitasvir/Paritaprevir/Ritonavir + Ribavirin (N=26) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir (N=210) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + Ribavirin (N=297)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hepatic Encephalopathy (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Drug Withdrawal Syndrome (General disorders) | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Abscess Limb (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Infected Cyst (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Alcohol Use (Social circumstances) | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/Ritonavir (N=1) | Ombitasvir/Paritaprevir/Ritonavir + Ribavirin (N=26) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir (N=210) | Ombitasvir/Paritaprevir/Ritonavir + Dasabuvir + Ribavirin (N=297)
Fatigue (General disorders) | 0 | 5 | 19 | 48
Headache (Nervous system disorders) | 0 | 3 | 13 | 33
Nausea (Gastrointestinal disorders) | 0 | 1 | 11 | 32
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 34
Insomnia (Psychiatric disorders) | 0 | 3 | 1 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT02581189/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT02581189/SAP_001.pdf